CLINICAL TRIAL: NCT02679833
Title: Effect of Toothpaste Fortified With Cyanocobalamin on Vitamin B12 Status: A 3 Month Placebo Controlled Randomized Study
Brief Title: Effect of Toothpaste Fortified With Cyanocobalamin on Vitamin B12 Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: Institute of Alternative and Sustainable Nutrition (IFANE) (Unknown)
Responsible Party: Principal Investigator, Rima Obeid, Prof. Dr., Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B12 status after toothpaste
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cobalamin Deficiency
Keywords: Cobalamin biomarkers; Anemia; Vegan diet; Subclinical; Metabolic functional markers; Holotranscobalamin; Methylmalonic acid
MeSH Terms: conditions — Vitamin B 12 Deficiency; Anemia | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A toothpaste, with the same matrix, all components, and appearance like the active arm but not containing vitamin B12.
  Interventions: Dietary Supplement: Placebo
- Cyanocobalamin (Active Comparator): A toothpaste with cyanocobalamin 100 µg cyanocobalamin per 1 g.
  Interventions: Dietary Supplement: Cyanocobalamin

INTERVENTIONS:
Dietary Supplement: Placebo — Toothpaste not containing the vitamin.
  Arms: Placebo
Dietary Supplement: Cyanocobalamin — Toothpaste containing100 µg cyanocobalamin/g.
  Arms: Cyanocobalamin

SUMMARY:
A 3 months randomized, placebo-controlled study on the effect of toothpaste fortified with vitamin B12 on vitamin B12 status markers and related metabolic markers. The primary outcome variable is the difference in the change of methylmalonic acid after 3 months between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Adults: men and women
* Stable diet for at least 24 months (omnivorous or a vegan diet).

Exclusion Criteria:

* Pregnancy and lactation
* Malabsorption disorders (Crohn disease, chronic gastritis, pernicious anemia, gastric or intestinal resection)
* Renal diseases
* Liver diseases
* Patients with cancer (or cancer history)
* Pre-study treatment with vitamin B12 or folate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The change in plasma concentrations of methylmalonic acid | Baseline, 3 months
  Lowering methylmalonic acid in the B12 arm compared with the placebo arm
The change in plasma concentrations of holotranscobalamin | Baseline, 3 months
  The effect on increasing holotranscobalamin in the B12 arm compared with the placebo arm
The change in plasma concentrations of homocysteine | Baseline, 3 months
  Lowering homocysteine in the B12 arm compared with the placebo arm
The change in plasma concentrations of vitamin B12 | Baseline, 3 months
  The effect on increasing plasma vitamin B12 in the B12 arm compared with the placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Markus Keller, PhD, Study Chair — Institute of Alternative and Sustainable Nutrition, Giessen, Germany; Rima Obeid, PhD, Study Director — Saarland University Hospital
Locations (2):
- Germany (2):
  - University of Saarland, Homburg, Saarland
  - Institute of Alternative and Sustainable Nutrition, Giessen

IPD SHARING:
Plan to Share IPD: No
Data sharing only between the two responsible study centers in a coded form, where participant ID is not shared.

REFERENCES:
- [Derived] Zant A, Awwad HM, Geisel J, Keller M, Obeid R. Vitamin B12-fortified toothpaste improves vitamin status in elderly people: a randomized, double-blind, placebo-controlled study. Aging Clin Exp Res. 2019 Dec;31(12):1817-1825. doi: 10.1007/s40520-019-01125-6. Epub 2019 Jan 24. PMID 30680547
- [Derived] Siebert AK, Obeid R, Weder S, Awwad HM, Sputtek A, Geisel J, Keller M. Vitamin B-12-fortified toothpaste improves vitamin status in vegans: a 12-wk randomized placebo-controlled study. Am J Clin Nutr. 2017 Mar;105(3):618-625. doi: 10.3945/ajcn.116.141978. Epub 2017 Jan 4. PMID 28052884